CLINICAL TRIAL: NCT06616493
Title: Tianjin University of Sport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin University of Sport (Other)
Responsible Party: Principal Investigator, Wei Zheng, Vice dean of school of exercise and health, Tianjin University of Sport, Tianjin University of Sport
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TJSport
Record Dates: First submitted 2024-09-22; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Effects of Kinesio Taping on Lower Extremity Biomechanical Characteristics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- KT (Experimental): subjects with kinesio taping
  Interventions: Other: kinesio taping
- placebo KT (Placebo Comparator): subjects with placebo kinesio taping
  Interventions: Other: kinesio taping
- control (No Intervention): subjects with no kinesio taping

INTERVENTIONS:
Other: kinesio taping — measure the subjects' lower extremity biomechanical characteristics with 3 different conditions respectively (kinesio taping, placebo kinesio taping, no taping)
  Arms: KT; placebo KT

SUMMARY:
Knee joint is one of the most important joints of the human body. It plays a vital role in basketball, football, volleyball and other sports that need to do repeated jumping and landing in high-speed sports. However, the rate of knee joint injury is high in sports, and knee joint injury often occurs in single leg landing. It is related to the decrease of flexion angle of hip and knee joint on the supporting side, the increase of extension and valgus moment, and the increase of ground reaction force. Kinesio taping has been widely used in the field of sports protection in recent years, but whether it can correct injury-related biomechanical risk factors is still controversial, and there are few studies on the timeliness changes of kinesio taping. Therefore, starting from the above concerns, this study compares the differences in biomechanical characteristics of lower limb joints in knee joints under three conditions : kinesio taping, placebo taping and no taping. At the same time, the changes of biomechanical characteristics of lower limbs before and after taping were observed in order to provide reference for the application of knee joint kinesio taping in sports injury protection.

ELIGIBILITY:
Inclusion Criteria:

* between 18-25 years old;
* BMI between 18.5-23.9kg/m2;
* no injury history or surgery history in recent six months.

Exclusion Criteria:

* kinesio taping allergy.

Ages: 21 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
hip flexion/extension angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  hip flexion/extension angle in sagittal plane at the initial touchdown moment
hip varus/valgus angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  hip varus/valgus angle in frontal plane at the initial touchdown moment
hip external/internal rotation angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  hip external/internal rotation angle in transverse plane at the initial touchdown moment
knee flexion/extension angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  knee flexion/extension angle in sagittal plane at the initial touchdown moment
knee varus/valgus angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  knee varus/valgus angle in frontal plane at the initial touchdown moment
knee external/internal rotation angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  knee external/internal rotation angle in transverse plane at the initial touchdown moment
ankle dorsiflexion/plantarflexion angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  ankle dorsiflexion/plantarflexion angle in sagittal plane at the initial touchdown moment
ankle varus/valgus angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  ankle varus/valgus angle in frontal plane at the initial touchdown moment
ankle external/internal rotation angle at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  ankle external/internal rotation angle in transverse plane at the initial touchdown moment
hip flexion/extension angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  hip flexion/extension angle in sagittal plane at the peak v-GRF moment
hip varus/valgus angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  hip varus/valgus angle in frontal plane at the peak v-GRFmoment
hip external/internal rotation angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  hip external/internal rotation angle in transverse plane at the peak v-GRF moment
knee varus/valgus angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  knee varus/valgus angle in frontal plane at the peak v-GRF moment
knee external/internal rotation angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  knee external/internal rotation angle in transverse plane at the peak v-GRF moment
knee flexion/extension angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  knee flexion/extension angle in sagittal plane at the peak v-GRF moment
ankle dorsiflexion/plantarflexion angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  ankle dorsiflexion/plantarflexion angle in sagittal plane at the peak v-GRF moment
ankle external/internal rotation angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  ankle external/internal rotation angle in transverse plane at the peak v-GRF moment
ankle varus/valgus angle at the peak vertical ground reaction force (v-GRF) moment | from enrollment to immediately after kinesio taping application
  ankle varus/valgus angle in frontal plane at the peak v-GRF moment
hip flexion/extension joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  hip flexion/extension joint torque in sagittal plane at the initial touchdown moment
hip varus/valgus joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  hip varus/valgus joint torque in the frontal plane at the initial touchdown moment
hip internal/external rotation joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  hip internal/external rotation joint torque in the transverse plane at the initial touchdown moment
knee flexion/extension joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  knee flexion/extension joint torque in sagittal plane at the initial touchdown moment
knee varus/valgus joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  knee varus/valgus joint torque in the frontal plane at the initial touchdown moment
knee internal/external rotation joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  knee internal/external rotation joint torque in the transverse plane at the initial touchdown moment
ankle dorsiflexion/plantarflexion joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  knee dorsiflexion/plantarflexion joint torque in sagittal plane at the initial touchdown moment
ankle varus/valgus joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  ankle varus/valgus joint torque in the frontal plane at the initial touchdown moment
ankle internal/external rotation joint torque at the initial touchdown moment | from enrollment to immediately after kinesio taping application
  ankle internal/external rotation joint torque in the transverse plane at the initial touchdown moment
hip flexion/extension joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  hip flexion/extension joint torque in sagittal plane at thepeak v-GRFmoment
hip varus/valgus joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  hip varus/valgus joint torque in the frontal plane at the peak v-GRF moment
hip internal/external rotation joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  hip internal/external rotation joint torque in the transverse plane at the peak v-GRF moment
knee flexion/extension joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  knee flexion/extension joint torque in sagittal plane at the peak v-GRF moment
knee varus/valgus joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  knee varus/valgus joint torque in the frontal plane at the peak v-GRF moment
knee internal/external rotation joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  knee internal/external rotation joint torque in the transverse plane at the peak v-GRF moment
ankle dorsiflexion/plantarflexion joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  ankle dorsiflexion/plantarflexion joint torque in sagittal plane at the peak v-GRF moment
ankle varus/valgus joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  ankle varus/valgus joint torque in the frontal plane at the peak v-GRF moment
ankle internal/external rotation joint torque at the peak v-GRF moment | from enrollment to immediately after kinesio taping application
  ankle internal/external rotation joint torque in the transverse plane at the peak v-GRF moment

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zheng, Study Director — Tianjin University of Sport, Tianjin, China
Locations (1):
- Wei Zheng, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided